CLINICAL TRIAL: NCT04680897
Title: Limits On Vaginal Intercourse After Mid-urEthral Sling (LOVE Trial)
Brief Title: LOVE Trial: Limits On Vaginal Intercourse After Mid-urEthral Sling
Acronym: LOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00070386
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Patient Satisfaction; Female Sexual Dysfunction
Keywords: mid-urethral sling
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The "early" group will be given instructions that allow them to return to vaginal penetration/intercourse after 2 weeks. The "standard" group will be given postoperative instructions that allow them to return to intercourse after 6 weeks. Both groups will be able to return to other physical activities as they feel able
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Other): Participants may resume vaginal penetration at 6 weeks.
  Interventions: Behavioral: Standard restriction recommendation
- Early Group (Other): Participants may resume intercourse at 2 weeks
  Interventions: Behavioral: Early restriction release

INTERVENTIONS:
Behavioral: Early restriction release — Participants will no longer have restrictions on vaginal penetration 2 weeks after surgery.
  Arms: Early Group
Behavioral: Standard restriction recommendation — Participants will return to intercourse after 6 weeks
  Arms: Standard Group

SUMMARY:
There are no prospective, randomized studies addressing vaginal penetration restrictions following mid-urethral slings. There is a single cohort study examining expedited recovery following vaginal prolapse repair which advised 3-weeks of vaginal penetration restrictions. This study reported an earlier return to intercourse in the 3-week group than in the retrospectively collected control group where 6-weeks of restriction were advised. This study did not evaluate the impact of early versus later return to sexual activity on wound complications, mesh exposure rates, pain or satisfaction.

It is important to develop evidenced-based recommendations on post-operative sexual activity restrictions.

The purpose of this research study is to understand if the "standard" 6-week restriction on vaginal penetration/intercourse after mid-urethral sling affects patient satisfaction

DETAILED DESCRIPTION:
The lifetime risk of surgery for stress urinary incontinence in women is 13.6%. Women are typically instructed to avoid strenuous physical activity and vaginal penetration for 6 weeks following synthetic mid-urethral sling procedures. The historical rationale behind these instructions was to prevent disruption of vaginal incisions, promote wound healing, decrease recurrence risk and prevent complications such as mesh exposure. Very little medical evidence exists, however, to support these activity restrictions which can have a negative impact on satisfaction and quality of life. Findings from a single randomized trial challenge standard activity restrictions following pelvic organ prolapse repair. Participants were given conservative or liberal postoperative instructions and the liberal group experienced fewer prolapse and urinary symptoms at 3 months postoperatively; but there was no difference in satisfaction between groups. This study, however, did not investigate restrictions on vaginal penetration (both groups adhered to 6-week restrictions) and was not specific to women undergoing isolated sling procedures. There are no prospective, randomized studies addressing vaginal penetration restrictions following mid-urethral slings. There is a single cohort study examining expedited recovery following vaginal prolapse repair which advised 3-weeks of vaginal penetration restrictions. This study reported an earlier return to intercourse in the 3-week group than in the retrospectively collected control group where 6-weeks of restriction were advised. This study did not evaluate the impact of early versus later return to sexual activity on wound complications, mesh exposure rates, pain or satisfaction.

Animal models suggest that wound healing occurs much sooner than 6 weeks post-surgery. In fact, epithelial wounds closed by primary intention typically re-epithelialize in just 24-48 hours. In a mouse-model with full-thickness vaginal injury, there was complete restoration of mucosal integrity by day 7 without surgical closure of the wound. Epithelial healing over mid-urethral sling could differ due to a known pro-inflammatory milieu in the setting of a mesh implant but the rate of epithelial closure over implanted synthetic mesh has not been specifically described. While earlier vaginal penetration could theoretically increase the risk of mesh exposure from the known baseline risk of 2-3%, this is unlikely following two weeks in a low risk population regardless of menopausal status. Vaginal atrophy has been identified as a risk factor for wound healing complications and vaginal mesh exposure and could interact with early resumption of intercourse. However, vaginal atrophy can be reversed with vaginal estrogen therapy and resultant risks mitigated.

Given the prevalence of mid-urethral slings for stress incontinence, it is important to develop evidenced-based recommendations on post-operative sexual activity restrictions. The purpose of this randomized trial, therefore, is to evaluate the impact of early (2 weeks) versus standard (6 weeks) removal of vaginal penetration restrictions in sexually active women undergoing mid-urethral sling procedures on sexual satisfaction and wound complications.

ELIGIBILITY:
Inclusion Criteria:

* At least 21years of age
* Women with stress or mixed urinary incontinence who are undergoing a planned, isolated, synthetic mid-urethral sling with cystoscopy via retropubic, transobturator or single-incision approach.
* Sexually active with ≥1 male or female partner with a frequency of at least once every 2 weeks
* Ability to comprehend the concept of randomization
* Willing to remain compliant with the instructions and study follow-up visits

Exclusion Criteria:

* History of prior surgery for incontinence including mid-urethral sling, fascial sling
* History of prior surgery for prolapse with transvaginal mesh
* Diabetic with Hgb A1C ≥ 8.0 % (elevated A1C is associated with delayed wound healing12 and 8.0 has been identified as a cutoff over which there are more complications postoperatively13
* Pregnant
* Incarcerated
* History of pelvic radiation
* Current smoker (known risk factor for mesh exposure)
* Non-English speaker

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender eligibility is not based on gender identity but on patients with female urethral anatomy.
Enrollment: 155 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction rating | week 12
  To determine if there is improved satisfaction with decreased length of restricted vaginal penetration following mid-urethral sling. The primary outcome will be patient satisfaction with ability to return to sexual function as measured on a 5-point Likert scale with the question: "How satisfied were you with your ability to return to vaginal penetration following surgery?"
  (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree

SECONDARY OUTCOMES:
Number of days until resumption of vaginal penetration | week 12
Number of Wound complications - wound separation | week 12
  To determine if there are increased wound complications in patients following isolated mid-urethral sling with shorter duration of restrictions on vaginal penetration.
Number of Wound complications - mesh exposure | week 12
  To determine if there are increased wound complications in patients following isolated mid-urethral sling with shorter duration of restrictions on vaginal penetration.
Number of Wound complications - mesh erosion | week 12
  To determine if there are increased wound complications in patients following isolated mid-urethral sling with shorter duration of restrictions on vaginal penetration.
Number of Wound complications - granulation tissue | week 12
  To determine if there are increased wound complications in patients following isolated mid-urethral sling with shorter duration of restrictions on vaginal penetration.
Number of Wound complications - vaginal pain | week 12
  To determine if there are increased wound complications in patients following isolated mid-urethral sling with shorter duration of restrictions on vaginal penetration.
Urinary incontinence | week 12
  To determine if there is similar continence in patients who resume intercourse early vs standard following isolated mid-urethral sling

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Matthews, MD, Principal Investigator — Wake Forest Health Sciences
Locations (3):
- United States (3):
  - Northwestern Medicine, Chicago, Illinois
  - Atrium Health, Charlotte, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04680897/ICF_000.pdf